CLINICAL TRIAL: NCT00477529
Title: A Phase I/II Trial of ABI-008 (Nab-docetaxel) in Patients With Hormone-refractory Prostate Cancer
Brief Title: ABI-008 Trial in Patients With Hormone-refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA301
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Hormone Refractory Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-008 (Experimental)
  Interventions: Drug: ABI-008

INTERVENTIONS:
Drug: ABI-008 — nab-docetaxel
  Other Names: nab-docetaxel

SUMMARY:
To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of ABI-008 given every 3 weeks; to characterize the toxicities of ABI-008; and to determine the pharmacokinetic parameters for ABI-008 when given on an every-3-week schedule.

DETAILED DESCRIPTION:
Detailed description not necessary.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study.

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate that is clinically refractory to hormone therapy.
2. Zubrod Performance Status 0-1.
3. At the time of enrollment, patients must have evidence of progressive metastatic disease, either:

   * Measurable disease with any level of serum PSA

     * OR
   * Non-measurable disease with PSA ≥ 5 ng/ml. Patients with PSA ≥ 5 ng/ml only and no other radiographic evidence of metastatic prostate cancer are not eligible.
4. Patients must have demonstrated evidence of progressive disease since the most recent change in therapy. Progressive disease is defined as any one of the following (measurable disease, bone scan, or PSA progression):

   * Measurable Disease Progression
   * Bone Scan Progression
   * PSA Progression
5. Serum testosterone ≤ 50 ng/ml, determined within two weeks prior to starting treatment.
6. Maintaining castrate status: Patients who have not undergone surgical orchiectomy should continue on medical therapies [e.g. gonadotropin releasing hormone analogs (GnRH analogs)] to maintain castrate levels of serum testosterone.
7. Megestrol acetate (MEGACE®) treatment may continue if patient has been on stable doses of the drug.
8. Age > 18 years of age.
9. Four weeks since major surgery.
10. The following restrictions on prior therapy for metastatic disease apply:

    * No prior chemotherapy regimen for metastatic disease.
    * No more than one prior course of palliative radiotherapy.
    * Up to one prior treatment with a non-chemotherapeutic agent (e.g., kinase inhibitors, immunotherapeutic agents, etc) is permitted as treatment for metastatic disease.
    * No prior radioisotope therapy with Strontium-89, Samarium or similar agents.
    * One prior neo-adjuvant or adjuvant chemotherapy regimen is permitted if given over 3 years ago.
11. No limitation on prior hormonal therapy.
12. Patients should be off all therapy for at least 4 weeks prior to study drug administration.
13. Life expectancy should be ≥ 3 months.
14. Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment.
15. Required Initial Laboratory Data:

    * WBC ≥ 3,000/µl
    * ANC ≥ 1,500/µl
    * Platelet count ≥ 100,000/µl
    * Creatinine ≤ 1.5 x
    * Total Bilirubin ≤ (exceptions will be made for patients with Gilbert's Disease)
    * SGOT (AST) ≤ 1.5 x
    * SGPT (ALT) ≤ 1.5 x
16. Men whose sexual partners are of child-bearing age must agree to use adequate contraception (hormonal or barrier method of birth control) for the duration of study participation.
17. If obese (weight > 20% of ideal body weight) patient must be treated with doses calculated using adjusted BSA.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study.

1. Patients may not be receiving any other investigational agents.
2. Patients may continue on a daily Multi-Vitamin, low dose (≤ 400 IU qd) Vitamin D, Calcitrol (≤ 0.5 mcg qd), and calcium supplements, but all other herbal, alternative and food supplements (i.e. PC-Spes, Saw Palmetto, St John Wort, etc.) must be discontinued before registration.
3. Patients on stable doses of bisphosphonates, who develop subsequent tumor progression, may continue on this medication.However, patients may not initiate bisphosphonate therapy prior to or during study
4. Patients with known brain metastases.
5. Patients with history of allergic reactions attributed to solvent-based docetaxel (Taxotere).
6. Patients with significant cardiovascular disease including congestive heart failure, active angina pectoris or recent myocardial infarction (within the last 6 months).
7. Patients with a "currently active" second malignancy other than non-melanoma skin cancers.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. HIV-positive patients receiving combination anti-retroviral therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2011-06-02 (Actual); Study Completion 2011-06-02 (Actual)

PRIMARY OUTCOMES:
DLT's and MTD's | 1 Year

SECONDARY OUTCOMES:
Efficacy of ABI-008 in this patient population | Q12 weeks and End of Study (EOS) and Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: John C Araujo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas